CLINICAL TRIAL: NCT05912881
Title: Chemosensory Dysfunction and Recovery in Endoscopic Endonasal Skull Base Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: North American Skull Base Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00311777
Record Dates: First submitted 2023-06-02; First posted 2023-06-22 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Anosmia; Skull Base Neoplasms
MeSH Terms: conditions — Anosmia; Skull Base Neoplasms | interventions — Olfactory Training

STUDY DESIGN:
Intervention Model Description: Participants are enrolled into treatment or placebo groups for the entirety of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study team members and study participants are blinded as to which olfactory training kit (treatment vs placebo) the participants received.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants receive placebo olfactory training kits that only contain medium chain triglycerides that lack any discernible odor
  Interventions: Other: Placebo training
- Treatment (Experimental): Participants receive treatment olfactory training kits that contain essential oils that have scents (lavender, lemon, clove, eucalyptus)
  Interventions: Other: Olfactory training

INTERVENTIONS:
Other: Olfactory training — Participants perform olfactory training using sticks filled with scented essential oils.
  Arms: Treatment
Other: Placebo training — Participants perform olfactory training using sticks filled with unscented medium chain triglycerides.
  Arms: Placebo

SUMMARY:
The investigators hypothesize that patients undergoing endoscopic endonasal skull base surgery experience clinically meaningful and modifiable disruptions in postoperative chemosensory function and quality of life, and the investigators further hypothesize that olfactory training in the postoperative period may significantly hasten normalization of patients' chemosensory perturbations. This tailored prospective study seeks to fulfill a significant gap in the understanding of the characteristics, implications, and treatment options for postoperative olfactory and gustatory impairment following endoscopic endonasal skull base surgery.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* preoperative diagnosis of benign sellar or parasellar skull base pathology

Exclusion Criteria:

* preoperative diagnosis of malignant sellar or parasellar skull base pathology
* history of endoscopic sinus surgery
* history of skull base surgery
* history of radiation therapy or other local treatments for the management of facial, sinonasal, or cranial pathologies
* history of chronic rhinosinusitis
* history of neurocognitive disorder
* history of intrinsic chemosensory pathology
* history of cardiac pacemaker
* history of gastrectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Olfactory function as assessed by the Sniffin Sticks olfactory testing kit | Pre-operative visit (baseline), 2 weeks post-operative, 1 month post-operative, 3 months post-operative
  Olfactory function as determined using the commercially available "Sniffin' Sticks" olfactory testing kit. Olfactory function is tested in three domains: threshold, discrimination, and identification. For threshold testing, the most dilute concentration of odorant that the participant is able to reliably detect is determined. In discrimination testing, the participant is evaluated on their ability to discern the unique scent among three scented sticks. In identification testing, the patient names the smells using a multiple choice form which offers four definitions for every Sniffin' stick, only one of which is correct.

SECONDARY OUTCOMES:
Change in Quality of Life as assessed by the Anterior Skull Base Nasal Inventory-12 | Pre-operative visit (baseline), 2 weeks post-operative, 1 month post-operative, 3 months post-operative, 6 months post-operative
  Quality of life questionnaire. Score range 0-60, where higher score is worse and indicates more onerous symptoms.
Change in Quality of Life as assessed by the ODOR (Olfactory Dysfunction Outcomes Rating) questionnaire | Pre-operative visit (baseline), 2 weeks post-operative, 1 month post-operative, 3 months post-operative, 6 months post-operative
  Quality of life questionnaire. Score range 0-112, where higher score is worse and indicates greater degree of olfactory dysfunction.
Change in Quality of Life as assessed by the Skull Base Inventory | Pre-operative visit (baseline), 2 weeks post-operative, 1 month post-operative, 3 months post-operative, 6 months post-operative
  Quality of life questionnaire. Score range 0-100, where higher score is better, indicative of less burden on quality of life.
Change in Quality of smell and taste as assessed by a Visual analog scale | Pre-operative visit (baseline), 2 weeks post-operative, 1 month post-operative, 3 months post-operative, 6 months post-operative
  Quality of smell and taste as indicated on a visual analog scale. Score range 0-100, where higher score is better and indicative of better smell and taste function.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Rowan, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Medicine, Baltimore, Maryland, United States